CLINICAL TRIAL: NCT02625649
Title: Effect of Gastric Bypass Surgery on Diabetes Status and Microvascular Complications in Obese Type 2 Diabetic Patients: Register-based and Clinical Follow-up Studies
Brief Title: Effect of Gastric Bypass Surgery on Diabetes Status and Microvascular Complications in Obese Type 2 Diabetic Patients
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 11092015
Record Dates: First submitted 2015-11-30; First posted 2015-12-09 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2016-10

CONDITIONS: Type 2 Diabetes Mellitus; Obesity; Diabetic Retinopathy; Diabetic Nephropathy
Keywords: Roux-en-Y gastric bypass; obesity; type 2 diabetes mellitus; diabetic nephropathy; diabetic retinopathy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetic Retinopathy; Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — blood samples urine samples stool samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RYGB: RYGB-operated type 2 diabetic patients
- non-RYGB: non-RYGB-operated type 2 diabetic controls

SUMMARY:
This study evaluates the long-term benefits of Roux-en-Y gastric bypass (RYGB) on type 2 diabetes mellitus, focussing on the prevalence and predictors of T2DM improvement and remission after RYGB, and subsequently relapse of type 2 diabetes mellitus after RYGB. Moreover, the study evaluates the possible effect of RYGB on diabetic microvascular complications such as nephropathy and retinopathy. Finally, the study provides insight into the factors influencing glucose-insulin homeostasis after RYGB, including altered microbiota diversity and bile acid levels.

DETAILED DESCRIPTION:
One hundred Danish type 2 diabetes mellitus (T2DM) patients who underwent Roux-en-Y gastric bypass surgery (RYGB) between 2006-2011 will be evaluated clinically together with 50 T2DM patients, matched on gender, age, presurgical body mass index, and diabetes duration.

The clinical follow-up consists of a physiological check-up, a thorough paraclinical work-up, and a whole body dual-energy x-ray absorptiometry (body composition and bone mineral density) a peripheral quantitative compute tomography (HR-pQCT), stool samples (microbiota), ophthalmological examination including retina photo, and a questionaire.

More over, a liquid meal test with sampling of total bile acids, fibroblast growth factor 19 and 21 (FGF 19 and FGF 21), plasma glucose, and insulin will be performed on a smaller part of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Capable
* type 2 diabetes mellitus
* speaks and understands Danish
* presents written concent
* cases must be Roux-en-Y operated between 2006-2011.

Exclusion Criteria:

* Converted Roux-en-Y
* chronic inflammatory bowel disease
* ischemic heart disease
* liver disease
* cholecystectomy.

Controls can not be bariatric operated.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Cases: Type 2 diabetes mellitus patients living in Central Denmark region that have undergone Roux-en-Y gastric bapass between 2006-2011.
  Controls: Type 2 diabetes mellitus patients living in Central Denmark region, non-RYGB-operated
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with HbA1c<48 mmol/mol. | Maximum follow-up is 121 months (january 2006-february 2016)

SECONDARY OUTCOMES:
Number of patients with T-score <-2,5 evaluated by dual energy xray absorptiometry | Maximum follow-up is 121 months (january 2006-february 2016)
Number of patients with urine albumin/creatinin< 30 mg/g | Maximum follow-up is 121 months (january 2006-february 2016)
Number of patients with two-step change from preoperative level on the Wisconsin Epidemiologic Study of Diabetic Retinopathy (WESDR) scale | From operation/inclusion to end of follow-up february 2016, maximum follow-up 121 months

CONTACTS AND LOCATIONS:
Overall Officials: Lene R Madsen, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Enodocrinology and Internal Medicine, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Madsen LR, Bek T, Richelsen B. Diabetic retinopathy in people with Type 2 diabetes and obesity treated by Roux-en-Y gastric bypass compared with non-operated controls: with focus on the role of diabetes remission in a cross-sectional and a 6-year follow-up study. Diabet Med. 2019 Apr;36(4):457-464. doi: 10.1111/dme.13876. Epub 2018 Dec 26. PMID 30537170